CLINICAL TRIAL: NCT06327074
Title: Feasibility Testing the Engaged Approach to Lung Cancer Screening
Brief Title: Testing the Engaged Approach to Lung Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-3063.cc
Record Dates: First submitted 2024-02-06; First posted 2024-03-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Sites in the control condition will be asked to complete appropriate/relevant surveys and interviews with minor modifications as needed and use the same Electronic Health Record Data Abstraction process.
- Experimental Group (Experimental): Sites randomized to use the EA-LCS materials will be given password-protected access to the program/toolkit web portal and encouraged to use any materials that fit the normal flow of clinic procedures. Materials available include both staff-facing and LCS candidate-facing materials.
  Interventions: Behavioral: Engaged Approach to Lung Cancer Screening

INTERVENTIONS:
Behavioral: Engaged Approach to Lung Cancer Screening — Sites randomized to use the EA-LCS materials will be given password-protected access to the program/toolkit web portal and encouraged to use any materials that fit the normal flow of clinic procedures. Materials available include both staff-facing and LCS candidate-facing materials.
  Staff-facing materials include:
  * Program website/manual/toolkit overview
  * Implementation insights with experts video series
  * Clinical placement placards
  * Program and clinician communication tools
  Candidate-facing materials include:
  * Program welcome letter
  * Maps and directions template
  * Communication preferences
  * Candidate letter templates (N=~8)
  * Program newsletter template and instructions
  * Lung nodule size comparison chart
  Other Names: EA-LCS
  Arms: Experimental Group

SUMMARY:
The goal of this study is to assess feasibility and acceptability of the Engaged Approach to Lung Cancer Screening (EA-LCS) in diverse lung cancer screening (LCS) programs operating in a variety of geographic regions across Colorado and the US.

ELIGIBILITY:
Inclusion Criteria:

The trial incorporates a multilevel assessment and enrollment involves inclusion criteria at two levels: (1) LCS Program and (2) LCS Program Staff member.

Program inclusion criteria (n = up to 8 sites):

* Must conduct at least 50 low-dose computed tomography (LDCT) scans per year (baseline + follow-up)
* Must be able to identify a primary contact person for LCS program operations (e.g., program coordinator, program navigator, program manager, etc.)

Staff member inclusion criteria (n ~ 5 at each site/~40 participants total):

* Identified staff member of the LCS program site
* >18 years of age
* Must be able to complete study surveys and interviews in English
* Willing to provide informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of the intervention group who would like to continue the EA-LCS framework | 7 months
Percentage of the intervention group who would recommend the EA-LCS framework to other programs | 7 months
Percentage of participants who would describe the framework as workable | 7 months

SECONDARY OUTCOMES:
Evaluate the intervention acceptability by Acceptability of Intervention Measure (AIM) | 12 months
  Indexes of intervention acceptability will be measured by the Acceptability of Intervention Measure (AIM).
  A 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean.
Evaluate the intervention appropriateness by Intervention Appropriateness Measure (IAM) | 12 months
  Indexes of intervention appropriateness will be measured by the Intervention Appropriateness Measure (IAM).
  A 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean.
Evaluate the intervention feasibility by Feasibility of Intervention Measure (FIM) | 12 months
  Indexes of intervention feasibility will be measured by the Feasibility of Intervention Measure (FIM).
  A 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Studts, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No